CLINICAL TRIAL: NCT06444256
Title: Orexin Receptor Antagonism and Sleep in Stimulant Use Disorder: A Pilot Study
Brief Title: Orexin Receptor Antagonism and Sleep in Stimulant Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Heather E. Webber, PhD, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0330
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Stimulant Use Disorder
Keywords: Psychostimulants; substance use; methamphetamine; cocaine
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SUVO (Experimental)
  Interventions: Drug: SUVO; Drug: TAU
- TAU (Active Comparator)
  Interventions: Drug: TAU

INTERVENTIONS:
Drug: SUVO — Participants will receive 20mg of SUVO for 7 days in the evening before bed on Day 5 through Day 11
  Arms: SUVO
Drug: TAU — Participants will receive supportive care and symptomatic medication per protocol at the inpatient facility.

SUMMARY:
The purpose of this study is to determine the effects of suvorexant (SUVO), on sleep, stress, and drug craving during early abstinence from stimulants and to determine the effects of treatment (SUVO vs. treatment as usual (TAU)) on post-treatment (Days 13-30) residential program length of stay (LOS) and completion rate.

ELIGIBILITY:
Inclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders(DSM-5)criteria for primary stimulant use disorder (either cocaine or methamphetamine)
* Be fluent in English and able to understand the consent form

Exclusion Criteria:

* Have an opioid use disorder of any severity
* Have a greater than moderate substance use disorder on any other substance
* Undergoing medication-assisted treatment for withdrawal of any substance
* Have any medical conditions contraindicating SUVO (e.g., severe pulmonary disease, severe cardiovascular disease or clinically abnormal ECG, severe liver or kidney disease, seizure disorder, or sleep disorder -particularly narcolepsy)
* Are currently taking medications with known drug interactions with SUVO (e.g., Monoamine oxidase (MAO) inhibitors, anticonvulsants, haloperidol, phenothiazines, anesthetics, and any sedative)
* Are pregnant or breast feeding
* BMI > 30 (women only)
* Have a current DSM-5 psychiatric disorder or neurological disease requiring on-going treatment that would make participation unsafe
* Have history of seizure disorder
* Have a head injury with loss of consciousness in the last 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in total sleep duration as assessed by the actigraphy watch | Baseline (Day 4), Day 5, day 6, day 7, day 8, day 9, day 10, day 11
Change in wake after sleep onset measured via actigraphy watch | Baseline (Day 4), Day 5, day 6, day 7, day 8, day 9, day 10, day 11
Change in self reported sleep quality as assessed by the Insomnia Severity Index (ISI) | Day 5 and Day 12
  This is a 7 item questionnaire and is rated on a five-point Likert scale ('0' representing none or not at all and '4' representing very much). Total scores range from 0 to 28, with higher combined scores indicating worse insomnia severity.
Changes in self reported sleep disturbance as assessed by the Patient Reported Outcomes Measurement Information System Short Form (PROMIS-SF) | Day 5 and Day 12
  This is a 4 item questionnaire and each is scored from 1-5 for a score range of 4-20, higher number indicating worse outcome
Changes in self reported Sleep-Related Impairment as assessed by the Patient Reported Outcomes Measurement Information System Short Form (PROMIS-SF) | Day 5 and Day 12
  This is an 8 item questionnaire and each is scored from 1-5 for a total score range of 8-40, higher number indicating worse outcome
Change in self-reported stress as assessed by the Visual Analog Scale (VAS) | Day 5 and Day 12
  This is measured from 0=no stress, 10=extreme stress
Change in stress and anxiety as assessed by the Depression, Anxiety and Stress Scale (DASS) | Day 5 and Day 12
  The DASS 21 is a 21 item self report questionnaire. Each item is scored from 0 (did not apply to me at all over the last week) to 3 (applied to me very much or most of the time over the past week), higher score indicating a worse outcome
Change in craving as assessed by the self reported Stimulant Craving Questionnaire (STCQ) | Day 5 and Day 12
  This is a 10 item questionnaire, each is scored from 0 (strongly disagree) to 6 (strongly agree) for a total score range of 0-60, higher score indicating worse outcome

SECONDARY OUTCOMES:
Change in resting state alpha power as assessed by EEG | Day 5 and Day 12
Change in stress as indicated by the amount of cortisol present in saliva during the cold-pressor task | Day 5 and Day 12
  Participants will submerge their hands in a bucket of ice water for up to 2 minutes and a saliva sample will be taken
Change in stress as indicated by the change in heart rate during the cold-pressor task | Day 5 and Day 12
  Participants will submerge their hands in a bucket of ice water for upto 2 minutes and heart rate will be measured
Change in stress as indicated by the change in systolic blood pressure during the cold-pressor task for upto 2 minutes | Day 5 and Day 12
  Participants will submerge their hands in a bucket of ice water for upto 2 minutes and blood pressure will be measured
Change in stress as indicated by the change in diastolic blood pressure during the cold-pressor task for upto 2 minutes | Day 5 and Day 12
  Participants will submerge their hands in a bucket of ice water for upto 2 minutes and blood pressure will be measured
Change in the amplitude of the Reward Positivity (RewP) component in microvolts in response to feedback on the Doors Task | Day 5 and Day 12
  The Doors Task will be used to elicit the RewP component, representing reward sensitivity. The task is a guessing game, where participants guess which door contains a reward behind it. After selecting a door, the participants are notified if they found the prize by a green arrow pointing up or if they did not find the prize by a red arrow pointing down.
Change in intensity of demand as assessed by the Drug Purchasing Task | Day 5 and Day 12
  Demand is the maximum quantity of Methamphetamine or Cocaine consumed if the drug was free measured in grams or dollar amount
Length of stay (LOS) | at time of discharge (up to 30 days form baseline)
Percentage of participants who complete the 30 day treatment | at time of discharge (up to 30 days form baseline)
Change in side effects as assessed by the side effects questionnaire | Day 5 , Day 12
  This 31-item questionnaire will be administered to assess side effects and adverse events in the SUVO group only

CONTACTS AND LOCATIONS:
Overall Officials: Heather Webber, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No